CLINICAL TRIAL: NCT03731663
Title: The Effect of Exposure to Food in Social Networks on Food Cravings and External Eating
Acronym: FEECAEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruppin Acdemic Center (Other)
Responsible Party: Principal Investigator, Efrat Neter, Associate Professor, Ruppin Acdemic Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 000000001
Record Dates: First submitted 2017-12-29; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Eating Habits and Behaviors, (UMLS)
Keywords: foodporn; food craving; external eating; disordered eating; social networks
MeSH Terms: conditions — Feeding Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: After receiving an explanation about the study and providing informed consent online, participants will complete questionnaires assessing demographic variables, SNS food preoccupation and disturbed eating online via Qualtrics link. Participants will then be randomly assigned to view a video clip showing pictures of either appetizing pictures of food (experimental group) or sightseeing pictures in a tourist destination (control group). After viewing the video, participants will respond to online questionnaire measuring external eating and food cravings, and will also be asked to order food they would like to eat immediately from a hypothetical menu.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appetizing Food exposure group (Experimental): Participants allocated to this group will watch a 3-minute video presenting a series of pictures of appetizing foods eaten in facilities in a tourist destination. An audio of a young adult describing herself eating these foods during a trip to London will be played.
  Interventions: Behavioral: Exposure to pictures of appetizing food (known as Foodporn)
- Control content watching group (Sham Comparator): Participants allocated to this group will watch a 3-minute video presenting a series of control pictures of tourist attractions in London. An audio of a young adult describing herself visiting these sites during a trip will be played.
  Interventions: Behavioral: Exposure to neutral pictures

INTERVENTIONS:
Behavioral: Exposure to pictures of appetizing food (known as Foodporn) — - Participants allocated to the experimental group will watch a 3 minute video presenting a series of pictures of appetizing foods. An audio of a young adult describing herself eating these foods during a trip to London will be played.
  Other Names: Experimental intervention
  Arms: Appetizing Food exposure group
Behavioral: Exposure to neutral pictures — Participants allocated to the control group will watch a 3 minute video presenting a series of control pictures of tourist attractions in London. An audio of a young adult describing herself visiting these sites during a trip will be played.
  Other Names: Control intervention
  Arms: Control content watching group

SUMMARY:
Background: Food practices are socially, culturally and historically embedded in everyday life. It is a common notion that people eat due to internal state of physiologic hunger but in fact the drive behind eating behaviors is much more complex. We eat, inter alia, because of our response to external cues such as the sight and smell of food, or external eating. Another related concept is food cravings: intense irresistible desires to consume a particular food that is distinct from hunger. Both external eating and food cravings have been associated with impulsivity, eating disorders and obesity. During recent decades the role of the media, and recently of the social media in our lives has grown significantly, and their influence on culture and society is now huge. A common activities on social media sites (SNS) is food viewing and posting pictures of tempting food, known as food porn. Food porn has been found to correlate with eating patterns and food-related attention and reward bias. The aim of this study is to conduct a controlled manipulation that may help us deduce causality as well as association. The investigators postulate that (1) viewing pictures of appetizing food will lead to higher rates of reported external eating and food craving than viewing pictures that are not food related; (2) Viewing these appetizing food pictures will lead participants to order different kinds of food and greater amounts; (3) The effect of viewing food pictures on external eating, food cravings and food orders will be greater for participants with high disturbed eating, then for participants without disturbed eating.

Method: After providing informed consent, 150 female participants (aged 18-35) will self report on demographic variables, SNS food preoccupation and disturbed eating (EAT-26). They will then be randomly assigned to watch either a food porn or control video. They will complete measures of food cravings (FCQ-S) and external eating (DEBQ) after watching the video and asked to order food they would like to eat from a virtual menu.)

DETAILED DESCRIPTION:
Participants Approximately 150 young participants (aged 18-35) will be recruited using a convenience sampling procedure. Participants will include Behavioral Science students at the Ruppin Academic Center who will be given credit points in exchange for participation on the stud, and young women recruited via social networks.

Measures Food cravings (state) will be assessed using the Food Craving Questionnaire (FCQ-S), a self report questionnaire with good psychometric properties (Cepeda-Benito, Gleaves, Willams, & Erath, 2000). The FCQ-S items are scaled on a five point Likret scale and measures five factors.

External eating will be assessed using the external eating scale in the Dutch Eating Behavior Questionnaire (DEBQ), a self-report questionnaire with good psychometric properties (van Strien, Frijters, Bergers, & Defares, 1986). The DEBQ measure restraint, emotional and external eating in different scales. The external eating scale contains ten statements scored on a five point Likret scale .

Disturbed eating will be assessed using the widely used Eating Attitude Test 26 (EAT-26) (Garner, Olmstead, Bohr, & Garfinkel, 1982). The EAT-26 is an 26-item measure of self reported symptoms and characteristics of EDs using a six point Likret scale (an example statement is "In the past 6 month have you: Exercised more than 60 minutes a day to lose or control your weight").

SNS food preoccupation will be measured by asking participant about specific food related SNSs activities and the frequency they engage in it. The activities include: frequency of posting food pictures on either Facebook or Instagram, frequency of encountering food pictures on either Facebook or Instagram, frequency of sending food pictures on WhatsApp, frequency of receiving food pictures on WhatsApp, frequency of following chefs, restaurants or brands on Instagram, frequency of posting pictures of food one prepared, frequency of posting pictures of food one is about to eat, frequency of taking pictures of ordered dishes in a restaurant, and lastly number of food-related groups one is a member of. The response on the first eighth questions was on a 5-point scale, ranging from 'never' to 'very often' and the response on the last question was on a 5-point scale, ranging from 0 to 7 and more. A total mean score of nine SNSs activities will be computed.

Design The independent variables will be the manipulated video (food versus non-food content), SNS use, SNS food preoccupation and disordered eating. External eating, food craving and food (type and amount) ordered will be the dependent variables.

Procedure After receiving an explanation about the study and providing informed consent online, participants will complete questionnaires assessing demographic variables, SNS food preoccupation and disturbed eating online via Qualtrics link. Participants will then be randomly assigned to view a video clip showing pictures of appetizing foods (experimental group) or neutral pictures of tourist destinations (control group). After viewing the video, participants will respond to online questionnaire measuring external eating and food cravings, and will also be asked to order food they would like to eat immediately from a hypothetical. The study will be approved by the IRB.

Statistical analyses Descriptive statistics will describe the characteristics of participants. Basic descriptive statistics will also be computed for the key variables of SNS use and eating patterns. The main analysis will examine the effect of the clip manipulation on external eating, food cravings and type and amount of food ordered, using MANCOVA, with disordered eating will be examined as a covariate. All statistical analyses will be performed using SPSS 23 (IBM SPSS Statistics, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

Age limits:

* Minimum (18), Unit of time (Years)
* Maximum (35) Unit of time (Years)
* Hebrew speaking, age 18-35

Exclusion Criteria:

* age (below 18 or over 35)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
External eating | Participants' external eating state will be measured immediately after the intervention. Up to 30 minuets after the end of intervention (The exact duration of questionnaire answering takes few minutes and varies between participants)
  External eating will be assessed using the external eating scale in the Dutch Eating Behavior Questionnaire (DEBQ), a self-report questionnaire with good psychometric properties. The DEBQ measure restraint, emotional and external eating in different scales. The external eating scale contains ten statements scored on a five point Likret scale.
Food cravings, state (situational) | Participants' food cravings state will be measured immediately after the intervention. Up to 30 minuets after the end of intervention (The exact duration of questionnaire answering takes few minutes and varies between participants).
  Food cravings (state) will be assessed using the Food Craving Questionnaire (FCQ-S), a self report questionnaire with good psychometric properties. The FCQ-S items are scaled on a five point Likret scale and measures five factors.
Type of ordered food | Up to 30 minuets after the end of intervention.
  Participants will be asked to order from a fixed menu the type of food they would like to eat immediately after the trial.
Amount of ordered food | Up to 30 minuets after the end of intervention.
  Participants will be asked to order from a fixed menu the amount of the chosen type of food they would like to eat immediately after the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruppin academic center, Emek Hefer, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bicen, H. (2015). Determination of University Students' Reasons of Using Social Networking Sites in their Daily Life. Procedia-Social and Behavioral Sciences, 190, 519-522. http://doi.org/10.1016/j.sbspro.2015.05.036
- [Background] Cepeda-Benito A, Gleaves DH, Fernandez MC, Vila J, Williams TL, Reynoso J. The development and validation of Spanish versions of the State and Trait Food Cravings Questionnaires. Behav Res Ther. 2000 Nov;38(11):1125-38. doi: 10.1016/s0005-7967(99)00141-2. PMID 11060941
- [Background] Coyne, S. M., Padilla-Walker, L. M., & Howard, E. (2013). Emerging in a digital world: A decade review of media use, effects, and gratifications in emerging adulthood. Emerging Adulthood, 1, 125-137.
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] McHale SM, Dotterer A, Kim JY. An Ecological Perspective on the Media and Youth Development. Am Behav Sci. 2009 Apr;52(8):1186-1203. doi: 10.1177/0002764209331541. PMID 22247564
- [Background] Mejova, Y., Abbar, S., & Haddadi, H. (2016). Fetishizing food in digital age:# foodporn around the world. Retrieved from http://arXiv preprint arXiv:1603.00229.
- [Background] Neely E, Walton M, Stephens C. Young people's food practices and social relationships. A thematic synthesis. Appetite. 2014 Nov;82:50-60. doi: 10.1016/j.appet.2014.07.005. Epub 2014 Jul 10. PMID 25017130
- [Background] Ruderman AJ. Dietary restraint: a theoretical and empirical review. Psychol Bull. 1986 Mar;99(2):247-62. No abstract available. PMID 3515384
- [Background] Santarossa, Sara, (2015)
- [Background] Schachter S, Goldman R, Gordon A. Effects of fear, food deprivation, and obesity on eating. J Pers Soc Psychol. 1968 Oct;10(2):91-7. doi: 10.1037/h0026284. No abstract available. PMID 5725907
- [Background] Spence C, Okajima K, Cheok AD, Petit O, Michel C. Eating with our eyes: From visual hunger to digital satiation. Brain Cogn. 2016 Dec;110:53-63. doi: 10.1016/j.bandc.2015.08.006. Epub 2015 Oct 1. PMID 26432045
- [Background] Van Strien, T., Frijters, J. E., Bergers, G., & Defares, P. B. (1986). The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International Journal of Eating Disorders, 5, 295-315.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03731663/Prot_SAP_000.pdf